CLINICAL TRIAL: NCT02863133
Title: Prospective, Multicenter, Multinational Study to Assess the Safety and Performance of the Easyx Antia Liquid Embolic in Intracranial Interventions IDEALE Study
Brief Title: Prospective Study to Assess the Safety and Performance of the Easyx Antia Liquid Embolic in Intracranial Interventions
Acronym: Ideale
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Antia Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 028
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Arterial Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Easyx Liquid Embolic (Experimental): embolization of intracranial malformations and fistulas and brain tumours with Easyx Liquid Embolic
  Interventions: Device: Liquid Embolic

INTERVENTIONS:
Device: Liquid Embolic — The Easyx liquid embolic, manufactured by Antia AG, is intended to occlude hypervascular lesions in the brain such as tumors, arteriovenous malformations (a tangle of abnormal and poorly formed blood vessels) and dural arteriovenous fistulas (abnormal connection of blood vessels).
  Other Names: Easyx

SUMMARY:
The study is a prospective, multicenter, multinational study to assess the safety and performance of the Easyx (trade name) Antia Liquid Embolic during embolization of intracranial malformations and fistulas. The clinical trial will include patients already scheduled for neuroradiological interventions. It is estimated that up to 8 sites will be required to collect the safety and performance data of the study material. Up to 65 patients will be enrolled in the study to achieve 53 evaluable patients. Each study centre will be required to treat 5 patients with a Dural arteriovenous fistula - DAVF before they can treat brain arteriovenous malformations - AVMs or brain tumours. Only experienced neuroradiologists will be invited to participate in this study.

DETAILED DESCRIPTION:
Study Procedures Once the subject has agreed to participate in the study and has signed the consent form, the baseline visit can be performed. A full medical history will be taken and a physical exam will be done as per local routine practice for an embolization procedure. The Cognard scale will be performed to assess the grade of a DAVF and the Spetzler Martin grade will be assessed if a brain AVM is to be treated; these are standard scoring systems for brain DAVFs and AVMs. A neurological exam will be done and any abnormalities will be documented.

Procedure Embolization of the DAVF or BAVM or tumor will be done as per routine practice but using the Easyx product. The procedure to treat a BAVM or a tumor may be staged and complex DAVFs may require a second treatment to fully occlude the fistula. The plan for treatment will be noted at the procedure visit and subsequent planned interventions will not be classed as adverse events. All interventions up to the 12 month follow up visit will be recorded in the Case Report Forms - CRFs. If the preliminary angiogram immediately prior to treatment shows that the target area can no longer be treated with an embolic product, the patient will be withdrawn from the study at this point and alternative treatment as per routine practice will be planned. Procedure details will be noted and feedback from the treating interventionalist will be collected, to determine the ease of handling of the product.

If the DAVF occlusion is complete, an assessment of where occlusion has been performed will be noted. If the DAVF or BAVM occlusion or blockage of the supply to a tumor is incomplete, the reason for incomplete occlusion will be given. The subject will be asked to complete a visual analog scale immediately after the procedure to report on any pain. A neurological exam will be done post treatment to assess for any changes.

Discharge The subject's condition will be recorded at discharge. Adverse events will be reported as well as any subsequent imaging or interventions that occurred following the initial treatment. A neurological exam will be done and any changes will be recorded. The Rankin score will only be done if there has been a hemorrhagic or ischemic stroke; this is a well known stroke scale.

One Month Follow up A follow up visit will be done at the clinic one month after the initial treatment. Adverse events will be reported and any subsequent imaging or interventions that occurred following the initial treatment. A neurological exam will be done and any changes will be recorded. The Rankin score will only be done if there has been a hemorrhagic or ischemic stroke.

Three - Six Months Follow up A control cerebral imaging will be done as per local routine practice for an embolization procedure. This may include dynamic Magnetic Resonance MR-Angiography, CT or catheter angiography. Adverse events will also be reported. The Cognard score and the Martin Spetzler grade will be documented and a neurological exam will be done. The Rankin score will only be done if there has been a hemorrhagic or ischemic stroke.

Twelve Months Follow up A final follow up visit will be done at 12 months to determine if any adverse events have occurred. A neurological exam will be done and any changes will be recorded. The Rankin score will only be done if there has been a hemorrhagic or ischemic stroke. Subjects may be brought back as late as 14 months post procedure, to fit in with routine follow up.

Risks

The clinical risks associated with the use of of Easyx™ and the procedure to place the device are the same as any other marketed embolic product. These risks of the procedure include:

* Headache
* Too much blood sugar
* Infection
* Bleeding from access point for delivery catheter
* Bleeding in the brain or a blood clot in the brain leading to stroke
* Low or high blood pressure
* Inability to get to the area to be treated
* Difficulty to remove the delivery catheter, entrapment of the catheter, rupture of the catheter
* Rupture of a blood vessel due to mishandling of the catheter or due to an attempt to free a catheter that has become stuck to the embolic agent
* Abnormal heart rhythm
* A tear in the wall of the blood vessel
* Respiratory failure
* Seizures
* Spasm of the blood vessels
* Fainting

The specific risks associated with the delivery of the embolic product itself are:

* Inability to clearly see the embolized area
* Allergic reaction related to placement of the embolic product
* Spasm of the blood vessels due to the solvent in the embolic product
* Low platelet count
* Reflux or migration of the embolic product
* Bleeding events related to product delivery
* Pain after the procedure, related to product delivery

The risks associated with the delivery system include:

* Catheter entrapment
* Catheter clogging
* Catheter rupture

The risks associated with the delivery of the embolic product into the incorrect target area are:

* Damage to the function of the cranial nerve vessels
* Symptoms of stroke associated with product being in the wrong brain vessels
* Tissue damage in the surrounding area of the embolic product
* Incorrect placement in the venous system

Benefits The liquid embolic EasyxTM has proved to be feasible and safe for endovascular embolization in animal AVM and hypervascular animal models. The main advantages of the material are its even consistency, strongly bound iodine providing high visibility under x-ray, the non stick properties in relation to the delivery catheter and the adhesive properties in relation to easy placement of the product in the target vessel. Also, the product is ready to use and so does not need any preparation prior to placement in the target vessel. These advantages show that Easyx is easy to use in comparison to other products already on the market. EasyxTM has been shown to be biocompatible. The solvent is quickly dispersed in the surrounding tissue allowing the embolic product to quickly precipitate in situ and provide a solid cast in a target vessel lumen.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 years or over
2. Subject exhibits a DAVF or BAVM or tumor that has been selected for endovascular treatment
3. Subject has provided written consent for the procedure.
4. Subject agrees to all follow up visits required by the protocol
5. The Subject is clinically and neurologically stable for a minimum of 48 hours prior to embolization.

Exclusion Criteria:

1. The subject has a brain AVM with high flow arteriovenous fistula that the investigator has determined to be unsuitable for embolization.
2. The subject has had acute cerebral bleeding within the last 6 months.
3. The patient is participating in another research study involving another investigational device, procedure or drug.
4. The brain AVM or DAVF or tumor has been previously treated with another embolization agent.
5. The subject has a bleeding disorder.
6. The subject is female and has a positive pregnancy test.
7. The subject has a life expectancy of less than 1 year.
8. Subject has a known allergy to contrast media used for radiography.
9. Subject has a known allergy to Dimethyl Sulfoxide - DMSO (solvent for the embolic product).
10. Subject has a condition that would prevent them attending follow up visits for up to 1 year.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Device related adverse events | 1 month
  The incidence of adverse events related to the device and procedure at 1 month follow up to ensure that the rate is equivalent to other products already on the market.
Technical Success | immediate
  The primary technical success endpoint is measured by evaluating the percentage achieved obliteration degree of the DAVF vascular lesion target or planned AVM region or vascular supply to a tumor. The assessment is done by means of a questionnaire

SECONDARY OUTCOMES:
Status of the lesion | 3 and 6 months
  Comparison of Cognard score (I, IIa, IIb, III, IV, V) for DAVFs and Spetzler Martin Grade (0, I, II, III, IV, V) for BAVMs pre and post treatment and at 3-6 months.The measures will be recorded in tables identifying and separating the scores
Useability | immediate
  Analysis of usability by a procedure questionnaire on the handling of the Easyx product
Neurological changes | 1, 6 and12 months
  A qualitative assessment if neurological changes appears at 1 month, 6 months and 12 months. If yes the changes will be itemized and described individually in a table

IPD SHARING:
Plan to Share IPD: Undecided